CLINICAL TRIAL: NCT01650142
Title: Study of the Neurofibromatosis 1 Expression: Identification of the Modifying Genes
Brief Title: Modifying Genes in Neurofibromatosis 1
Acronym: NFGENMODIF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French National Referral Center for Neurofibromatoses (Unknown)
Responsible Party: Sponsor
Other Study IDs: AOM 10 005; 2010-023137-34 (EudraCT Number)
Record Dates: First submitted 2012-05-29; First posted 2012-07-26 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Neurofibromatosis 1
Keywords: Neurofibromatosis 1; Phenotype; Modifiers
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NF1GeneModif Cohort: Adult patients with neurofibromatosis 1
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Thanks to the investigators previous study the investigators demonstrated the influence of modifying genes in the phenotypic expression of neurofibromatosis 1 (Hum Mol Genet. 2009; 18 (15) :2768-78). Indeed, analysis of the intra-and inter-family variability performed using the investigators phenotype/genotype database demonstrated a strong genetic component for most clinical features. The investigators results suggest the involvement of genetic factors, not related to the NF1 gene, the modifiers. The objective of this project is to identify the modifiers involved in the variability of clinical expression of NF1. The investigators will focus in particular variants involved in the development and progression of neurofibromas.

DETAILED DESCRIPTION:
Neurofibromatosis 1(NF1) is a rare autosomal dominant disorder with an incidence of one birth out of 3000. NF1 gene is located in 17q11.2. The penetrance is near 100% by the age of 8 and the de novo mutations represent half the cases. The product of NF1 gene is neurofibromin, a protein controlling cellular differentiation and proliferation. Phenotypic expression is variable even in the same family. Neurofibromatosis 1 is characterized by café au lait spots, freckling of the folds, Lisch'nodules (hamartomas of iris) and multiple neurofibromas. Manifestations of neurofibromatosis 1 are pleiotropic, potentially severe and unpredictable. Morbidity and mortality associated to neurofibromatosis 1 are linked with complications, optic pathway gliomas, neurofibromas of the spine or of peripheral nerves, learning disabilities, scoliosis and bone abnormalities and vasculopathy. The investigators already demonstrated the existence of modifiers, genes modifying the phenotypic expression of neurofibromatosis 1 (Hum Mol Genet. 2009;18(15):2768-78). Indeed, a quantitative analysis of inter and intrafamilial variability performed with the data of the investigators phenotype/genotype database showed a strong genetic component for most studied clinical traits with an estimated heritability from 44 and 45% for subcutaneous and plexiform neurofibromas, to 66% for small café au lait spots. The investigators also showed that the NF1 gene had minor effect in the phenotypic variability. The investigators results suggested the implication of genes non linked to NF1 gene. The identification of these variants called modifiers of the phenotype is possible thanks to the investigators vast collection of patients and its statistical power. The aim of the present study is to identify in the human genome genetic variants in the evolving pattern of the most frequent manifestation of neurofibromatosis 1, neurofibromas. The genetic association studies are the most adapted in that purpose. The investigators bank includes at the present time 1099 patients of 575 families with genotypes, phenotypes and DNA samples.

The investigators will include 450 index cases more to have around 1000 independent patients with neurofibromatosis 1 to get a 90% statistical power to detect variants of 30% frequency in the general population and having an effect of odds ratio of 2 for studied trait. The investigators will use Affymetrix® Genechips 6.0 covering well the whole genome.

Identification of the variants will provide new comprehension of pathophysiology and new targets for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged of 18 or more
* Patient with neurofibromatosis 1 according the NIH criteria :
* Six or more café au lait macules over 15 mm in greatest diameter in postpubertal individuals
* Two or more neurofibromas of any type or one plexiform neurofibroma
* Freckling in the axillary or inguinal regions (Crowe´s sign)
* Optic glioma
* Two or more Lisch nodules (iris hamartomas)
* A distinctive osseous lesion such as sphenoid dysplasia or thinning of long bone cortex with or without pseudoarthrosis
* A first-degree relative (parent, sibling, or offspring) with NF1 by the above criteria
* The criteria are met in an individual if two or more of the features listed are present.

Exclusion Criteria:

* Children (< 18 year-old)
* One member of the family already included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with neurofibromatosis 1 according to the NIH criteria followed in NF France network, a national network devoted in to neurofibromatosis 1
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Identification of the genetic variants involved in variability of clinical expression of neurofibromatosis 1. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Wolkenstein, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Easton DF, Ponder MA, Huson SM, Ponder BA. An analysis of variation in expression of neurofibromatosis (NF) type 1 (NF1): evidence for modifying genes. Am J Hum Genet. 1993 Aug;53(2):305-13. PMID 8328449
- [Background] Gutmann DH, Aylsworth A, Carey JC, Korf B, Marks J, Pyeritz RE, Rubenstein A, Viskochil D. The diagnostic evaluation and multidisciplinary management of neurofibromatosis 1 and neurofibromatosis 2. JAMA. 1997 Jul 2;278(1):51-7. PMID 9207339
- [Background] Sabbagh A, Pasmant E, Laurendeau I, Parfait B, Barbarot S, Guillot B, Combemale P, Ferkal S, Vidaud M, Aubourg P, Vidaud D, Wolkenstein P; members of the NF France Network. Unravelling the genetic basis of variable clinical expression in neurofibromatosis 1. Hum Mol Genet. 2009 Aug 1;18(15):2768-78. doi: 10.1093/hmg/ddp212. Epub 2009 May 5. PMID 19417008